CLINICAL TRIAL: NCT06542484
Title: The Real-world Treatment Satisfaction by Gefapixiant in Patients with Refractory Chronic Cough in Terms of Cough Improvement and Taste Disturbance. (The RESTORE Study)
Brief Title: The Real-world Treatment Satisfaction by Gefapixiant in RCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nagoya City University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Yoshihiro Kanemitsu, Lecturer, Nagoya City University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NagoyaCU-RCC
Record Dates: First submitted 2024-08-05; First posted 2024-08-07 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-12

CONDITIONS: Chronic Cough
Keywords: Chronic Cough; gefapixiant
MeSH Terms: conditions — Chronic Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gefapixiant arm (Experimental): Participants will take 45mg of gefapixiant twice a day for 12 weeks.
  Interventions: Drug: Gefapixant Citrate

INTERVENTIONS:
Drug: Gefapixant Citrate — An additional treatment of gefapixiant will be performed for 12 weeks.
  Other Names: LYFNUA Tablets

SUMMARY:
Chronic cough has a high global prevalence and it is refractory to such treatments by approximately 20% of patients. Gafapixant is a P2X3 receptor antagonist that has demonstrated the reduction of cough in patients with refractory chronic cough(RCC). Taste disturbance is the most frequent adverse event by gefapixant (approximately 60-70%). Although gefapixant is well-tolerated even if taste disturbance has occurred, the impact of taste disturbance on cough-specific QoL remains to be unclear. Therefore, the investigator would like to evaluate factors related to treatment satisfaction by gefapixant in RCC patients. the investigator hypothesize that taste disturbance will be associated with the improvement of cough specific QoL and treatment satisfaction in RCC patients.

DETAILED DESCRIPTION:
Chronic cough has a high global prevalence, but appears to be poorly recognized. Most patients respond to specific treatments against causes of chronic cough. Meanwhile, cough is refractory to such treatments by approximately 20% of patients and they are regarded as "refractory chronic cough (RCC). Gafapixant is a P2X3 receptor antagonist that has demonstrated the reduction of cough in patients with RCC through the inhibition of ATP transmission to afferent nerves. According to the COUGH-1 and COUGH-2, taste disturbance is the most frequent adverse event by gefapixant, with the incidence of 59.3% in COUGH-1 and 68.9% in COUGH-2, respectively. Although 45 mg of gefapixant is well-tolerated even if taste disturbance has occurred, the impact of taste disturbance on cough-specific QoL remains to be unclear in RCC and UCC. Furthermore, both taste disturbance and the improvement of cough by gefapixant would be associated with treatment satisfaction. Therefore, the investigator would like to evaluate factors related to treatment satisfaction by gefapixant in RCC patients. The investigator hypothesize that taste disturbance will be associated with the improvement of cough specific QoL and treatment satisfaction in RCC patients. Furthermore, the investigator would like to evaluate the association of taste disturbance with cough-specific QoL in the real-world clinical practice. In addition, there are no biomarkers available that can predict the efficacy of the improvement of cough by gefapixant. The investigator will also explore biomarkers that can be helpful in predicting well response to gefapixant in RCC and UCC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with RCC and UCC (8 weeks or more).
2. Cough is refractory to intensive specific treatments for causes of chronic cough.
3. Never smokers and ex-smokers with having smoking history of ≤20 pack-years.

Exclusion Criteria:

1. Patients with lung cancer, interstitial lung diseases, bronchiectasis, or respiratory infection such as tuberculosis and acute pneumonia.
2. Current smoker, ex-smokers with having smoking history of >20 pack-years, or those who quit smoking within six months prior to receiving gefapixant.
3. Those who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Treatment satisfaction | 12 weeks
  To evaluate the change in treatment satisfaction with the initiation of gefapixiant and to determine factors related to treatment satisfaction by gefapixant. The investigator will assess overall treatment satisfaction using 5-point Likert scale (1. Very dissatisfied 2. Dissatisfied 3. Neutral 4. Satisfied 5. Very Satisfied) at enrolment and 12 weeks after commencing gefapixant from all participants. The investigator will compare the rate of "Satisfaction" (4. Satisfied 5. Very Satisfied) before and after the initiation of gefapixant using the McNemar analysis. Taste disturbance will also be assessed using the Patient-Reported Outcome version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) classification with slight modification (Grade 0: No change in taste. Grade 1: Altered taste but no change in diet, Grade 2: Altered taste with change in diet; noxious or unpleasant taste; loss of taste; Grade 3 Cease to gefapixant due to altered taste)

SECONDARY OUTCOMES:
The change in cough-specific quality of life and clinical factors | 12 weeks
  To evaluate the association between the change in cough-specific quality of life (QoL) using the Leicester Cough Questionnaire (LCQ) and the change in clinical factors with gefapixant. The LCQ questionnaire consists of 19 items with 3 domains. It ranges from 3 to 21, with higher scores indicate better cough-specific QoL.
The changes in the core five tastes | 12 weeks
  To evaluate the changes in the core five tastes such as sweet, sour, bitter, salty, and umami with the initiation of gefapixiant and to determine what tastes are associated with the change in cough-specific quality of life (QoL). The investigator will evaluate threshold of five basic taste perception with a whole-mouth method using a series of twofold dilutions of the taste solutions including sweet (sucrose), salty (NaCl), sour (tartaric acid), bitter (quinine HCl), and umami (monosodium L-glutamate). These measurements will be conducted before and 12 weeks after the initiation of gefapixant to investigate which taste will be affected by gefapixant. The investigator will prepare for 8 doubling concentrations of these 5 tastes, respectively. Sucrose, citric acid, NaCl, Munosodium glutamate, and quinine HCL will be used to make solutions.
Seeking biomarkers | 12 weeks
  To seek biomarkers that can predict the change of cough-specific quality of life by gefapixant. Lack of zinc and copper are well-known cause of taste disturbance. Copper/zinc ratio is reported as a good diagnostic marker for taste disorders. Thus, the investigator thinks that they may be associated with the development of taste disturbance by gefapixant. The investigator will measure them because their levels will be helpful when considering the additional zinc therapy for taste disorder in clinical practice. The investigator will also use airway immune cells obtained from sputum samples to measure the expression CD 39 and CD 73 in sputum.

CONTACTS AND LOCATIONS:
Overall Officials: Yoshihiro Kanemitsu, Principal Investigator — Nagoya City University Graduate School of Medical Sciences and Medical School
Locations (2):
- Japan (2):
  - Nagoya City University, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken

IPD SHARING:
Plan to Share IPD: No